CLINICAL TRIAL: NCT00452634
Title: A Phase II Study of Irinotecan/Cisplatin Plus Simvastatin in Chemo-naive Patients With Extensive Disease-Small Cell Lung Cancer
Brief Title: Irinotecan/Cisplatin Plus Simvastatin in Extensive Disease-Small Cell Lung Cancer (ED-SCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Ji-youn Han, Head of Lung Cancer Center, National Cancer Center, Korea
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-06-176
Record Dates: First submitted 2007-03-26; First posted 2007-03-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Small Cell Lung Cancer
Keywords: Irinotecan; cisplatin; Simvastatin; Extensive disease; SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Irinotecan; Cisplatin; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- study arm (Experimental)
  Interventions: Drug: Irinotecan; Drug: Cisplatin; Drug: Simvastatin

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 65mg/m2/iv over 90min on day 1 and 8, repeat Q 3weeks. until disease progression, unacceptable toxicity or patients' refusal.
Drug: Cisplatin — Cisplatin 30mg/m2/iv over 30min on day 1 and 8, repeat Q 3weeks. until disease progression, unacceptable toxicity or patients' refusal.
Drug: Simvastatin — simvastatin 40mg/QD, PO, daily, every 3 weeks

SUMMARY:
3-Hydroxy-3-methylglutaryl CoA reductase inhibitors, commonly referred to as the statins, have proven therapeutic and preventative effects in cardiovascular diseases. Recently, there are emerging interests in their use as anticancer agents based on preclinical evidence of their antiproliferative, proapoptotic, anti-invasive, and radiosensitizing properties. Inhibition of 3-hydroxy-3-methylglutaryl CoA reductase by the statins interferes with the rate-limiting step of the mevalonate pathway, leading to reduced levels of mevalonate and its downstream products, many of which play important roles in critical cellular functions such as membrane integrity, cell signaling, protein synthesis, and cell cycle progression. Perturbations of these processes in neoplastic cells by the statins may therefore result in control of tumor initiation, growth, and metastasis. The statins have demonstrated growth inhibitory activity in cancer cell lines and preclinical tumor models in animals. Simvastatin, a member of the statin family, profoundly impaired basal and growth factor-stimulated SCLC cell growth in vitro and induced apoptosis. SCLC cells treated with simvastatin were sensitized to the effects of the chemotherapeutic agent etoposide. Moreover, SCLC tumour growth in vivo was inhibited by simvastatin. Therefore, the investigators will conduct this phase II trial to evaluate the efficacy & toxicity of irinotecan/cisplatin plus simvastatin in patients with chemo-naïve ED-SCLC.

DETAILED DESCRIPTION:
Cisplatin-30 mg/m2 on day 1 and 8 repeat q 3 weeks Irinotecan-65 mg/m2 on day1 and 8 repeat q 3 weeks Simvastatin 40 mg per day orally from D1 of cycle 1

Treatment will be continued until disease progression, unacceptable toxicity, or patients' refusal.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of SCLC
* Extensive-stage disease, defined as disease extending beyond one hemithorax or involving contralateral mediastinal, hilar or supraclavicular lymph nodes, and/or pleural effusion.
* No prior chemotherapy, immunotherapy, or radiotherapy
* Performance status of 0, 1, 2 on the ECOG criteria.
* At least one unidimensional measurable lesion meeting Response Evaluation Criteria in Solid Tumors (RECIST. 2000).
* Patient compliance that allow adequate follow-up.
* Adequate hematologic (WBC count ≥ 4,000/mm3, platelet count ≥ 150,000/mm3), hepatic (bilirubin level ≤ 1.5 mg/dL, AST/ALT ≤ 80 IU/L), and renal (creatinine concentration ≤ 1.5 mg/dL) function.
* Informed consent from patient or patient's relative.
* Males or females at least 18 years of age.
* If female: childbearing potential either terminated by surgery, radiation, or menopause, or attenuated by use of an approved contraceptive method (intrauterine device [IUD], birth control pills, or barrier device) during and for 3 months after trial. If male, use of an approved contraceptive method during the study and 3 months afterwards. Females with childbearing potential must have a urine negative HCG test within 7 days prior to the study enrollment.
* No concomitant prescriptions including cyclosporin A, valproic acid, phenobarbital, phenytoin, ketoconazole.
* Patients with brain metastasis are allowed unless there were clinically significant neurological symptoms or signs

Exclusion Criteria:

* Inability to comply with protocol or study procedures.
* A serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* A serious cardiac condition, such as myocardial infarction within 6 months, angina, or heart disease, as defined by the New York Heart Association Class III or IV.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrollment.
* Concurrent administration of any other antitumor therapy.
* Pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2006-04; Primary Completion 2009-11 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
1-year survival & overall survival | the first day of treatment to death or last survival confirm date

SECONDARY OUTCOMES:
Tumor response rate | the ratio between the number of responders and number of patients assessable for tumor response
Time to progression | the first day of treatment to the date that disease progression is reported
Toxicity | the first date of treatment to 30 days after the last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Youn Han, M.D.,Ph.D., Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyenggi, South Korea